CLINICAL TRIAL: NCT03722186
Title: An Open-label, Single-arm, Phase I Study of the Safety, Tolerability and Pharmacokinetic/Pharmacodynamic Characteristics of SHR-1603 in Subjects With Advanced Solid Tumor or Relapsed/Refractory Lymphoma
Brief Title: Safety, Tolerability and Pharmacokinetics/Pharmacodynamics (PK/PD) of SHR-1603 in Subjects With Advanced Malignancies
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1603-I-101
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Physiological Effects of Drugs; Neoplasms by Histologic Type; Lymphoma; Hematologic Neoplasms; Immunotherapy; Advanced Cancer
Keywords: advanced solid tumor; R/R lymphoma
MeSH Terms: conditions — Neoplasms by Histologic Type; Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1603 (Experimental): Multiple escalating doses of SHR-1603
  Interventions: Drug: SHR-1603

INTERVENTIONS:
Drug: SHR-1603 — SHR-1603 monotherapy

SUMMARY:
SHR-1603-I-101 is an single-arm, open-label, dose finding phase I clinical trial of SHR-1603 in subjects with advanced solid tumor or relapsed/refractory malignant lymphoid diseases. The study drug will be administered by intravenous infusion.

DETAILED DESCRIPTION:
SHR-1603-I-101 is a single-arm, open-label, dose finding, first-in-human(FIH) clinical trial of SHR-1603 intravenous infusion in subjects with advanced solid tumor or relapsed/refractory malignant lymphoid diseases.

The primary objective of this study is to evaluate the safety and tolerability of SHR-1603, as well as to determine the maximally tolerated dose(MTD) and define the recommended Phase 2 dose(RP2D) of SHR-1603.

The study is consisted of a dose-escalation Part 1 followed by a dose expansion Part 2 and a clinical expansion Part 3.

Part 1 will use accelerated titration and 3+3 dose-escalation design to determine MTD.

Part 2 will further evaluate the safety, tolerability and PK/PD features of SHR-1603 based on the results of Part 1.

Part 3 will include several cohorts of malignancies to collect preliminary efficacy information of SHR-1603.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years or older;
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
3. Life expectancy no less than 12 weeks;
4. Pathologically confirmed advanced solid tumor or relapsed/refractory lymphoma with measurable target lesions;
5. Adequate bone marrow, haptic, renal and coagulation function.

Exclusion Criteria:

1. Evidence of central nervous system (CNS) involvement;
2. Previously treated with similar agents;
3. History of anticancer treatment within 4 weeks of enrollment (6 weeks for subjects treated with nitrosoureas or mitomycins);
4. Anticipated to be involved in other anti-cancer treatments expect for palliative care during the trial;
5. History of anti-cancer vaccination; or history of vaccination using attenuated vaccines within 4 weeks of enrollment;
6. History of Red blood cell (RBC) transfusion within or treatment with erythropoitin(EPO) within 3 months of enrollment;
7. History of grade 3 or higher thrombolic incidence within 2 years of enrollment, or using antithrombotic/anticoagulant agents;
8. With confirmed immunodeficiency, uncontrolled auto-immune disease, uncontrolled cardiovascular disease, uncontrolled or active infection;
9. Substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events(AE) of SHR-1603 | 18 months (anticipated)
  Assessment of the incidence of treatment-emergent AEs
Dose-limited toxicity (DLT) of SHR-1603 | 18 months(anticipated)
  Assessment of the incidence of DLT
Maximum tolerated dose (MTD) of SHR-1603 | 18 months(anticipated)
  The highest dosing level at which no more than 1 of 6 patients has DLT

SECONDARY OUTCOMES:
The peak plasma concentration (Cmax) of SHR-1603 | 18 months (anticipated)
  The serum concentrations of SHR-1603 at each dose level, between the first and second intravenous administration.
The area under the plasma concentration versus time curve (AUC) of SHR-1603 | 18 months (anticipated)
  The plot of SHR-1603 concentration in blood plasma versus time after intravenous infusion.
The half-life(t1/2) of SHR-1603 | 18 months (anticipated)
  The time required for the serum concentration of SHR-1603 be reduced to half of its peak concentration.
The objective response rate(ORR) in subjects with advanced tumors treated with SHR-1603 | 36 months
  The proportion of patients with reduction in tumor burden. RECIST 1.1(solid tumor) or LUGANO 2014(lymphoma) will be used for assessment.
The best of response (BOR) in subjects with advanced tumors treated with SHR-1603 | 36 months
  The best response recorded from the start of the study treatment until the disease progression. RECIST 1.1(solid tumor) or LUGANO 2014(lymphoma) will be used for assessment.
The progression free survival (PFS) in subjects with advanced tumors treated with SHR-1603 | 36 months
  Time from the first dose of SHR-1603 until disease progression or death. Disease progression will be determined according to RECIST 1.1(solid tumor) or LUGANO 2014(lymphoma).
The Duration of response (DoR) in subjects with advanced tumors treated with SHR-1603 | 36 months
  Time from documentation of tumor response to disease progression. RECIST 1.1(solid tumor) or LUGANO 2014(lymphoma) will be used for assessment.
The disease control rate (DCR) in subjects with advanced tumors treated with SHR-1603 | 36 months
  The percentage of subjects with solid tumor who have achieved complete response(CR), partial response(PR) and stable disease(SD) no less than 24 weeks since start of treatment. RECIST 1.1(solid tumor) or LUGANO 2014(lymphoma) will be used for assessment.
The clinical benefit rate (CBR) in subjects with advanced tumors treated with SHR-1603 | 36 months
  The percentage of subjects with solid tumor who have achieved complete response(CR), partial response(PR) and stable disease(SD). RECIST 1.1(solid tumor) or LUGANO 2014(lymphoma) will be used for assessment.
SHR-1603 receptor occupation | 30 months
  red blood cell and white blood cell surface receptor occupation will be assessed frequently
SHR-1603 antibodies | 30 months
  anti SHR-1603 antibodies will be tested frequently

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No